CLINICAL TRIAL: NCT01828255
Title: A Single Center, Case-control, Open Label Study Assessing Intraocular Pressure Patterns in Patients With Primary Open-angle Glaucoma Experiencing Fast Versus Slow Visual Field Progression
Brief Title: Intraocular Pressure (IOP) Patterns in Fast Versus Slow Visual Field (VF) Progression Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1212
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Primary Open-angle Glaucoma (POAG) Patient
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish® (Experimental): Device: portable device that monitors the 24-hour IOP pattern by a wireless contact lens sensor placed on the eye that sends its signals via an antenna around the orbital cavity to a recorder. Upon completion, the recording can be transmitted to a computer for read-out and visualization.
  Interventions: Device: SENSIMED Triggerfish®

INTERVENTIONS:
Device: SENSIMED Triggerfish®

SUMMARY:
The purpose of this study is to investigate how the intraocular pressure (IOP) varies in time and if the IOP variations are associated with the worsening of glaucoma. IOP patterns will be recorded continuously over 24 hours with SENSIMED Triggerfish® (TF) a portable investigational device using a contact lens sensor. After completing the Triggerfish lens placement and removal; the patient will complete a formal Polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 89 years old
* Diagnosis of treated POAG (including normal tension glaucoma (NTG))
* All IOP measurements during the VF period (to be described further) equal or lower than 18 mmHg and/or on average equal or lower than 16 mmHg in the same period
* Documented glaucomatous VF damage at baseline, characterized by glaucoma hemifield test result outside normal limits on at least 2 consecutive VF tests or the presence of at least 3 contiguous test points within the same hemifield on the pattern deviation plot at p<0.01, with at least 1 point at p < 0.005
* At least 8 visual field tests carried out within at least 2 years, all with fixation losses and false positive/negative results equal or less than 33%
* For fast progressing eyes, 1) pointwise progression defined as two or more adjacent VF test locations in the same hemifield that show a threshold sensitivity rate of change more negative than -1.0 dB/year with p<0.01 or 2) a global rate of VF change based on mean deviation (MD) more negative than -1.0 dB/year
* For slowly or minimally progressing eyes a VF MD rate of change more positive than -0.5 dB/year with no significant pointwise progression as described above
* Not more than 6 diopters spherical equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Baseline VF MD more negative than -15 dB. The rationale here is that in severely damaged visual fields, one may not be able to detect and measure rates of progression due to a 'floor effect'
* Corneal or conjunctival abnormality precluding contact lens adaptation
* Severe dry eye syndrome or other ocular disease
* Patients with angle closure glaucoma, traumatic glaucoma or uveitic glaucoma
* Patients with previous intraocular surgery in the enrolled eye, including cataract surgery
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in unrelated clinical research within the last 4 weeks

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo De Moraes, MD, Principal Investigator — The New York Eye and Ear Infirmary; Jeffrey M Liebmann, MD, Principal Investigator — The New York Eye and Ear Infirmary; Robert Ritch, MD, Principal Investigator — The New York Eye and Ear Infirmary
Locations (1):
- The New York Eye and Ear Infirmary, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fast Progressors: pointwise progression defined as two or more adjacent VF test locations in the same hemifield that show a threshold sensitivity rate of change more negative than -1.0 dB/year with p<0.01 or a global rate of VF change based on MD more negative than -1.0 dB/year
- Slow Progressors: VF MD rate of change more positive than -0.5 dB/year with no significant point defined as two or more adjacent VF test locations in the same hemifield that show a threshold sensitivity rate of change more negative than -1.0 dB/year with p<0.01wise progression
Period: Overall Study
Arm/Group | Fast Progressors | Slow Progressors
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Slow Progressors: VF MD rate of change more positive than -0.5 dB/year with no significant pointwise progression defined as two or more adjacent VF test locations in the same hemifield
- Total: Total of all reporting groups
Arm/Group | Slow Progressors | Fast Progressors | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.3) | 68.3 (8.6) | 67 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Visual field defect [Mean (Standard Deviation); unit: dB] — Visual field is measured by perimetry and the mean defect (MD) is assesses the defect in the visual field.
  dB | -0.07 (0.12) | -1.88 (0.48) | -0.98 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between 24-hour IOP Pattern as Recorded by TF and VF Progression in Patients With POAG.
Description: 24-hour measurement of TF, corresponding to IOP-related fluctuations expressed in arbitrary units of mini volts equivalent (mVeq) and comparison of this measurement between POAG patients showing fast and slow rates of glaucoma visual field progression.
Time Frame: 24-hour
Population: POAG patients with slow or fast rate of VF glaucoma progression
Measure: Mean (Standard Deviation); unit: mVeq
Groups:
- Fast Progressors: Patients with a fast rate of progression (<-1dB/y)
- Slow Progressors: Patients with a slow rate of progression (>-1dB/y)
Arm/Group | Fast Progressors | Slow Progressors
Number analyzed (Participants) | 17 | 17
mVeq | 410.1 (138.4) | 334.6 (119.4)

2. Secondary Outcome: Relationship Between TF Pattern and VF Progression According to TF Slope
Description: Measurement of TF, corresponding to IOP-related fluctuations expressed in arbitrary units of mini volts equivalent (mVeq) and comparison of this measurement between POAG patients showing fast and slow rates of glaucoma visual field progression during wake vs sleep periods. The wake slope corresponds to the change in the TF signal from 1 hour before to 1 hour after the time the subject went to sleep. The sleep slope corresponds to the change from 1 hour before to 1 hour after the time the subject awoke.
Time Frame: 24-hour
Population: POAG patients with slow or fast rate of VF glaucoma progression
Measure: Mean (Standard Deviation); unit: mVeq/hour
Groups:
- Fast: Pointwise progression defined as two or more adjacent VF test locations in the same hemifield that show a threshold sensitivity rate of change more negative than -1.0 dB/year with p<0.01 or a global rate of VF change based on MD more negative than -1.0 dB/year
- Slow: VF MD rate of change more positive than -0.5 dB/year with no significant pointwise progression defined as two or more adjacent VF test locations in the same hemifield
Arm/Group | Fast | Slow
Number analyzed (Participants) | 17 | 17
mVeq/hour
  Wake slope | 34.9 (55.7) | 34.6 (44.3)
  Sleep slope | -33.5 (44.6) | -35.7 (61.9)

3. Secondary Outcome: Relationship Between TF Pattern and VF Progression According to Day and Night
Description: TF measurement during diurnal and nocturnal periods and comparison of this measurement between POAG patients showing fast and slow rates of glaucoma visual field progression.
Time Frame: 24-hour
Measure: Mean (Standard Deviation); unit: mVeq
Arm/Group | Fast | Slow
Number analyzed (Participants) | 17 | 17
mVeq
  Diurnal | 84.0 (37.2) | 93.9 (40.6)
  Nocturnal | 30.8 (9.6) | 42.3 (16.0)

4. Secondary Outcome: Relationship Between 24-hour TF Pattern and VF Progression According to TF Peak
Description: Number of peaks in 24-Hours TF pattern, defined as the local maximum point in the smoothed TF profile.
Time Frame: 24-hour
Measure: Mean (Standard Deviation); unit: Number of peaks
Arm/Group | Fast | Slow
Number analyzed (Participants) | 17 | 17
Number of peaks | 13.1 (3.0) | 14.1 (4.9)
Statistical Analysis 1: Comparison: Fast vs Slow; Test type: Other; p < 0.005, t-test, 2 sided

5. Secondary Outcome: 24-hour TF IOP Pattern in Patients With POAG With Fast and Slow Rates of VF Progression
Description: Comparison (Spearman correlations) between 24-hour IOP-related fluctuations measured by TF and 24-hour blood pressure profiles (systolic, diastolic and mean arterial blood pressure) of POAG patients showing fast and slow rates of glaucoma visual field progression. The correlation between TF and blood pressure measurement was calculated within each subject then mean values were obtained for patients with slow vs fast glaucoma visual field progression.
Time Frame: 24-hour
Measure: Mean (Standard Deviation); unit: coefficient of correlation
Arm/Group | Fast | Slow
Number analyzed (Participants) | 17 | 17
coefficient of correlation
  Systolic blood pressure | -0.08 (0.32) | -0.19 (0.32)
  Diastolic blood pressure | -0.06 (0.36) | -0.22 (0.30)
  Mean arterial blood pressure | -0.06 (0.35) | -0.21 (0.28)

ADVERSE EVENTS:
Arm/Group | Fast Progressors | Slow Progressors
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fast Progressors (N=20) | Slow Progressors (N=20)
Corneal abrasion (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No